CLINICAL TRIAL: NCT06713122
Title: The Effect of Symptom Management Training Given to Gynaecological Cancer Patients Receiving Chemotherapy With Artificial Intelligence Supported Mobile Application on Supportive Care Needs, Symptom Severity and Psychological Well-Being
Brief Title: Effects of Symptom Management Education With Mobile Application in Gynecological Cancer Patients Receiving Chemotherapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Esra Nur Erdoğan (Other)
Responsible Party: Sponsor-Investigator, Esra Nur Erdoğan, Associate Investigator, PhD Student, Research Assistant, Saglik Bilimleri Universitesi
Organization: Saglik Bilimleri Universitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-442
Record Dates: First submitted 2024-11-10; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-12

CONDITIONS: Gynaecological Cancer; Chemotherapy; Nursing Care
Keywords: Gynaecological cancer; chemotherapy; mobile application; nursing care; psychological well-being; supportive care needs
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group- Group receiving Symptom Management Training with Mobile Application (Experimental): Mobile application intervention will be applied to the intervention group. The evaluation tests will be repeated after the first cycle of chemotherapy treatment, at the 3rd and 5th cycles.
  Interventions: Behavioral: İntervention Group- Group receiving Symptom Management Training with Mobile Application
- Control Group (No Intervention): No intervention will be applied to the control group. The evaluation tests will be repeated after the first cycle of chemotherapy treatment, at the 3rd and 5th cycles.

INTERVENTIONS:
Behavioral: İntervention Group- Group receiving Symptom Management Training with Mobile Application — The application to be developed in the research will be both Android and IOS supported.
  Monitoring the active use of the patients from the interface by the researcher and receiving individual and collective notifications in line with the profile that the patients receiving chemotherapy will create in the application will increase the usability of the application. Thus, the benefit that users receive after active use can be determined.
  The content of the Let's fight the symptoms together module will be created by experts in the field and people will be able to actively use these methods while struggling with the symptoms they experience.
  Patients may not always have the opportunity to reach a nurse or health professional. In symptom management with the mobile application, artificial intelligence will be trained by the researcher and integrated into the application will help patients reach the right information without wasting time.
  Arms: İntervention Group- Group receiving Symptom Management Training with Mobile Application

SUMMARY:
Gynaecological cancers, which have an important place among the cancers seen both in the world and in our country. Chemotherapy, which is one of the most commonly used and basic methods in cancer treatment, causes many physical and psychological side effects while treating the disease. It is very important to identify the symptoms experienced, evaluate, control and provide professional health guidance.

The spread of digitalisation has turned mobile learning into a kind of need or necessity rather than a preference. Increases the control of individuals over themselves and provides self-discipline.

The aim of this study was to evaluate the effect of symptom management training given with an artificial intelligence supported mobile application on supportive care needs, symptom severity and psychological well-being of gynaecological cancer patients receiving chemotherapy.

The study was planned as a randomised controlled trial. The population of the study will consist of patients who applied to Etlik City Hospital-Oncology Hospital-Day Outpatient Unit for the first time to receive chemotherapy treatment for gynaecological cancer and completed the first course.

The study will be conducted with a total of 70 patients, including 35 patients from the intervention group and 35 patients from the control group.

Research Hypotheses:

Gynaecological cancer patients receiving chemotherapyBetween the intervention group receiving symptom management training with a mobile application and the control group receiving standard care;

1. H1: There is a difference in terms of the severity of symptoms experienced.
2. H2: There is a difference in terms of supportive care needs.
3. H3: There is a difference in terms of psychological well-being levels. Data Collection Tools Descriptive Information Form, Edmonton Symptom Diagnostic Scale, Supportive Care Needs Scale, Psychological Well-Being Scale and Eastern Cooperative Oncology Group (ECOG) Performance Scale will be used as data collection tools.

Modules to be included in the Mobile Application:

The forms will be administered a total of three times, initially at the end of the 3rd and 5th cycle.

Module 1: Introducing Module Module 2: Application Usage Instruction Module Module 3: Recognise the Disease Module Module 4: Common Symptoms and Recommendations During Chemotherapy Treatment Module Module 5: Let's Fight Symptoms Together Module Module 6: Ask Anything - Counselling Module

DETAILED DESCRIPTION:
Gynaecological cancers, which have an important place among the cancers seen both in the world and in our country, are malignant tumours of the female reproductive organ. In the treatment of gynaecological cancers, many methods such as chemotherapy, radiotherapy, surgical treatment, hormone therapy are used alone or together. Chemotherapy, which is one of the most commonly used and basic methods in cancer treatment, causes many physical and psychological side effects while treating the disease. However, side effects may not occur at the same time and some may develop after discharge. Therefore, it is very important to identify the symptoms experienced, evaluate, control and provide professional health guidance.

The spread of digitalisation has turned mobile learning into a kind of need or necessity rather than a preference. The use of web-based platforms in disease management leads to effective communication between the patient and the healthcare team. Thanks to the use of a web-based platform, communication between the patient and the caregiver increases, saving time and reducing costs. In addition to the benefits such as the ability of the health professional to plan the treatment planning by incorporating the patient's experiences, needs and concerns into the process and providing the benefit of access without spatial limitations, it also increases the control of individuals over themselves and provides self-discipline.

The aim of this study is to evaluate the effect of symptom management training given with an artificial intelligence supported mobile application developed for gynaecological cancer patients receiving chemotherapy on supportive care needs, symptom severity and psychological well-being.

The study was planned as a randomised controlled trial. Block randomisation will be used to assign patients to intervention and control groups.

The population of the study will consist of patients who applied to Etlik City Hospital-Oncology Hospital-Day Outpatient Unit for the first time to receive chemotherapy treatment for gynaecological cancer and completed the first course.

The sample of the study will consist of patients who applied to Etlik City Hospital-Oncology Hospital-Day Outpatient Unit to receive chemotherapy treatment for the first time and who meet the following inclusion criteria.

The study will be conducted with a total of 70 patients, including 35 patients from the intervention group and 35 patients from the control group (The sample number of the study was calculated by using the G Power programme using the data of a study in which mobile application intervention was carried out on cancer patients. Accordingly, the confidence interval was 95%; the margin of error was accepted as 5% and a total of 56 patients were found as 28 intervention and 28 control group. Considering that there may be losses during the mobile application intervention, the sample number was kept 25% higher than the calculated sample number.)

Research Hypotheses:

Gynaecological cancer patients receiving chemotherapyBetween the intervention group receiving symptom management training with a mobile application and the control group receiving standard care;

1. H1: There is a difference in terms of the severity of symptoms experienced.
2. H2: There is a difference in terms of supportive care needs.
3. H3: There is a difference in terms of psychological well-being levels. Data Collection Tools Descriptive Information Form, Edmonton Symptom Diagnostic Scale, Supportive Care Needs Scale, Psychological Well-Being Scale and Eastern Cooperative Oncology Group (ECOG) Performance Scale will be used as data collection tools.

   * Data collection tools will be sent to patients via the application and will be asked to be filled in.

Modules to be included in the Mobile Application:

* The application will include module, registration, login and profile creation sections.
* The intervention group will be able to give feedback as they use the application.
* Motivational messages will be sent.
* At the end of the study, the mobile application will also be open to the control group.
* The forms will be administered a total of three times, initially at the end of the 3rd and 5th cycle.
* Module 1: Introducing Module
* Module 2: Application Usage Instruction Module
* Module 3: Recognise the Disease Module
* Module 4: Common Symptoms and Recommendations During Chemotherapy Treatment Module
* Module 5: Let's Fight Symptoms Together Module
* Module 6: Ask Anything - Counselling Module

ELIGIBILITY:
Inclusion Criteria:

* Receiving chemotherapy for the first time due to gynaecological cancer and completing the first chemotherapy course
* At least 18 years old
* Not previously diagnosed with cancer, diagnosed with gynaecological cancer for the first time and only
* Literate
* Who agreed to participate in the research
* No communication barrier
* Eastern Cooperative Oncology Group (ECOG) Performance Scale score below 3
* No diagnosed psychiatric illness
* Women who have an Android or IOS smartphone and can access the internet

Exclusion Criteria:

* The investigator discontinued the treatment
* Chemotherapy treatment discontinued after the start of the study
* Not actively using the mobile application
* Not filling in the forms during the use of the Mobile Application
* The occurrence of another cancer during the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Supportive Care Needs | Evaluation test: will be performed after the first cycle of chemotherapy treatment and after the 3rd and 5th cycles (each cycle is 28 days)
  Supportive Care Needs Scale:Each question in the scale is numbered from 1 to 5 and 1 point corresponds to 'I did not experience this situation' and 5 points correspond to 'I needed a lot of support'
Symptom Severity | Evaluation test: will be performed after the first cycle of chemotherapy treatment and after the 3rd and 5th cycles (each cycle is 28 days)
  Edmonton Symptom Diagnostic Scale: The severity of each symptom is assessed with numerical numbers from 0 to 10. A score of 0 indicates that the symptom is absent and a score of 10 indicates that the symptom is felt very severely.
Psychological Well-Being | Evaluation test: will be performed after the first cycle of chemotherapy treatment and after the 3rd and 5th cycles (each cycle is 28 days)
  Psychological Well-Being Scale: The items of the Psychological Well-Being Scale are answered between 1-7 in the form of strongly disagree (1) and strongly agree (7). Scores vary between 8 and 56. A high score indicates that the person has many psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Esra Nur Erdoğan, PhD Student, Study Chair — University of Health Sciences Gulhane Faculty of Nursing, Department of Obstetrics and Gynaecology; Gülten Güvenç, Prof.Dr., Principal Investigator — University of Health Sciences Gulhane Faculty of Nursing, Department of Obstetrics and Gynaecology; Tülay Eren, Asst. Prof., Study Chair — Etlik City Hospital, Medical Oncology
Locations (1):
- Etlik City Hospital-Oncology Hospital-Day Outpatient Unit, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After the end of the study: study protocol and Clinical Study Report (CSR)
Supporting Information: Study Protocol, CSR
Time Frame: After the end of the study

REFERENCES:
- [Background] Graetz I, Anderson JN, McKillop CN, Stepanski EJ, Paladino AJ, Tillmanns TD. Use of a web-based app to improve postoperative outcomes for patients receiving gynecological oncology care: A randomized controlled feasibility trial. Gynecol Oncol. 2018 Aug;150(2):311-317. doi: 10.1016/j.ygyno.2018.06.007. Epub 2018 Jun 11. PMID 29903391

DOCUMENTS (3):
  • Study Protocol (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT06713122/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT06713122/SAP_001.pdf
  • Informed Consent Form (2024-09-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT06713122/ICF_002.pdf